CLINICAL TRIAL: NCT03112161
Title: The Effects of Energy Imbalance on Food Intake Behaviors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 05-0067; R01DK072174 (NIH)
Record Dates: First submitted 2017-04-07; First posted 2017-04-13 (Actual); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Eucaloric (Experimental): Participants will consume a eucaloric diet with a macronutrient composition of 20% protein, 30% fat and 50% carbohydrate for 4 days (Eucaloric Feeding Period). The caloric value of the diet will be calculated based on lean body mass plus an activity factor to ensure energy and macronutrient balance.
  Interventions: Other: Eucaloric Feeding Period
- Overfed (Experimental): Following 3 days of eucaloric feeding, participants will complete a 1-day overfeeding period (Overfeeding Feeding Period), during which their diet will have a daily energy value of 40% greater than the eucaloric diet (Eucaloric Arm), although the macronutrient composition will remain the same (20% protein, 30% fat, 50% carbohydrate).
  Interventions: Other: Overfeeding Feeding Period
- Underfed (Experimental): Following 3 days of eucaloric feeding, participants will complete a 1-day underfeeding period (Underfeeding Feeding Period), during which their diet will have a daily energy value of 40% less than the eucaloric diet (Eucaloric Arm), although the macronutrient composition will remain the same (20% protein, 30% fat, 50% carbohydrate).
  Interventions: Other: Underfeeding Feeding Period

INTERVENTIONS:
Other: Eucaloric Feeding Period
  Arms: Eucaloric
Other: Overfeeding Feeding Period
  Arms: Overfed
Other: Underfeeding Feeding Period
  Arms: Underfed

SUMMARY:
This study will determine whether changes in energy balance alter regional neuronal activation of brain regions associated with food intake in individuals screened to be either resistant or prone to obesity. Specifically, it will determine whether foods of "hedonic" value elicit changes in regional neuronal activity in the fasted and fed state in "obese-resistant" and "obese-prone" men and women in varying states of energy balance.

ELIGIBILITY:
Inclusion Criteria:

In the obese-prone group:

* BMI between 20-30
* Report at least one obese first-degree relative
* Self-describe as "struggling" with weight
* Weight-stable for at least 3 months prior to study participation

In the obese-resistant group:

* BMI between 17-25
* Report no obese first-degree relatives
* Self-describe as "naturally thin" and have never been overweight
* Overall weight stability

Exclusion Criteria:

* Significant medical or psychiatric disease
* History of eating disorder
* Left handed
* Unable to complete an MRI scan (e.g., metal in body, claustrophobic)

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2005-06-14 (Actual); Primary Completion 2015-10-01 (Actual); Study Completion 2015-10-01 (Actual)

PRIMARY OUTCOMES:
Change in neuronal response to food vs. nonfood objects in fasted vs. fed states | Day 5 of each of the three 5-day study periods (Eucaloric, Overfeeding, Underfeeding)
  Change in neuronal response to food vs. nonfood objects in the overfed and underfed feeding periods as compared to the eucaloric period between fasted and fed states in obese-prone as compared to obese-resistant individuals.

SECONDARY OUTCOMES:
Change in appetite ratings | At baseline, in the fasted state on Day 5 of each of the three 5-day study periods (Eucaloric, Overfeeding, Underfeeding) and at 30, 90, 120, 150 and 180 minutes after a meal on Day 5 of each of the three 5-day study periods.
  Change in appetite ratings via visual analog scale (VAS; 0-100) before vs. after a meal in the overfeeding and underfeeding periods compared to the eucaloric feeding periods between obese-resistant and obese-prone individuals.
Change in food cravings | At baseline and both before and after a meal on Day 5 of each of the three 5-day study periods (Eucaloric, Overfeeding, Underfeeding).
  Change in food cravings (questionnaire) before vs. after a meal in the overfeeding and underfeeding periods compared to the eucaloric feeding periods between obese-resistant and obese-prone individuals.
Change in leptin levels | At baseline, in the fasted state on Day 5 of each of the three 5-day study periods (Eucaloric, Overfeeding, Underfeeding) and at 30, 90, 120, 150 and 180 minutes after a meal on Day 5 of each of the three 5-day study periods.
  Change in blood leptin levels before vs. after a meal in the overfeeding and underfeeding periods compared to the eucaloric feeding periods between obese-resistant and obese-prone individuals.
Change in ghrelin levels | At baseline, in the fasted state on Day 5 of each of the three 5-day study periods (Eucaloric, Overfeeding, Underfeeding) and at 30, 90, 120, 150 and 180 minutes after a meal on Day 5 of each of the three 5-day study periods.
  Change in blood ghrelin levels before vs. after a meal in the overfeeding and underfeeding periods compared to the eucaloric feeding periods between obese-resistant and obese-prone individuals.
Change in PYY levels | At baseline, in the fasted state on Day 5 of each of the three 5-day study periods (Eucaloric, Overfeeding, Underfeeding) and at 30, 90, 120, 150 and 180 minutes after a meal on Day 5 of each of the three 5-day study periods.
  Change in blood Peptide YY (PYY) levels before vs. after a meal in the overfeeding and underfeeding periods compared to the eucaloric feeding periods between obese-resistant and obese-prone individuals.
Change in neuronal response to hedonic vs. basic food images | Day 5 of each of the three 5-day study periods (Eucaloric, Overfeeding, Underfeeding)
  Change in neuronal response to hedonic vs. basic food images in the overfed and underfed feeding periods as compared to the eucaloric period between fasted and fed states in obese-prone as compared to obese-resistant individuals.
Change in body weight | Baseline and every 6 months for up to 5 years after study participation.
  Change in body weight from baseline for up to 5 years in obese-resistant and obese-prone individuals

CONTACTS AND LOCATIONS:
Overall Officials: Jason Tregellas, PhD, Principal Investigator — University of Colorado, Denver; Marc-Andre Cornier, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No